CLINICAL TRIAL: NCT03904966
Title: The Effect of Low-dye Kinesio Taping in Addition to Extracorporeal Shock Wave Therapy in Patients With Plantar Fasciitis
Brief Title: The Effect of Kinesio-tape and Shock Wave Therapy on Plantar Fasciitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hitit University (Other)
Responsible Party: Principal Investigator, Yeliz Bahar Ozdemir, Principal Investigator, Hitit University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19KAEK063
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Plantar Fascitis; Calcaneus Spur
MeSH Terms: conditions — Heel Spur | interventions — Athletic Tape; Extracorporeal Shockwave Therapy

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Outcomes Assessor
Masking Description: To ensure group concealment, randomization will be done by using opaque, sealed envelopes and the assessors will be blinded to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ESWT+ Kinesiotaping (Experimental): Low-dye Kinesio taping technique 4 times in 5 weeks in addition to extracorporeal shock wave therapy
  Interventions: Device: Kinesio tape; Device: Extracorporeal shock wave therapy
- ESWT+Shamtaping (Sham Comparator): Sham taping technique 4 times in 5 weeks in addition to extracorporeal shock wave therapy
  Interventions: Device: Kinesio tape; Device: Extracorporeal shock wave therapy
- ESWT (Other): Extracorporeal shock wave therapy for 5 sessions (5-week)
  Interventions: Device: Extracorporeal shock wave therapy

INTERVENTIONS:
Device: Kinesio tape — Kinesio tape will be applied on the plantar heel (the most painful area) of the patients for the treatment of plantar fasciitis, in addition to the extracorporeal shock wave therapy
  Arms: ESWT+ Kinesiotaping; ESWT+Shamtaping
Device: Extracorporeal shock wave therapy — Extracorporeal shock wave therapy will be used for all patients with plantar fasciitis. (5 sessions for 5-week)

SUMMARY:
Foot problems are common in society. Accordingly, loss of workforce, quality of life and mental health deterioration can be observed in employees and hardship in daily life activities, balance-walking problems and fall risk increase in older adults. The presence of athletic and sedentary populations causes a large number of patients to apply to outpatient clinics with the complaint of heel pain every year. Plantar fasciitis (plantar heel pain), although multifactorial origin, obesity, overload bearing and ankle joint motion reduction factors are thought to play an active role in the emergence of discomfort.

Foot orthoses are a common treatment used for plantar heel pain, but a period of several weeks is usually required between the diagnosis and transportation to the orthosis due to the production process. Therefore, short-term therapies such as supportive banding are used to alleviate the symptoms of this intermediate period. The low-dye taping technique is the most commonly used banding technique and has been found to be effective in randomized controlled trials. In addition, there is a rare study in the literature showing the efficacy of Kinesio taping method. Although both were found to be useful in the treatment of plantar fasciitis, no randomized controlled trial was studied in this patient population of the low-dye method with Kinesio taping. In the studies, the early period of banding therapy is mentioned and studies on relatively longer treatment response are still required. Our hypothesis is that low-dye Kinesio-banding treatment added to ESWT treatment for patients diagnosed with plantar fasciitis will be effective on foot functionality by reducing the pain of the patient both in the early and later period.

DETAILED DESCRIPTION:
One of the most common musculoskeletal pathologies of the foot and pain is plantar heel pain. In the studies, it was stated that the feeling of foot pain and stiffness was between 18% and 63%. The plantar fascia is the most common cause of heel pain in adult age. Due to overuse, such as standing for a long time or running, it is assumed that it occurs as a result of micro-injury on the surface of the plantar fascia. It has been reported that 10% of the general population will be encountered throughout life. Although the exact cause is not known, middle age, obesity, excessive foot pronation, pes cavus, running, pes planus and long-term standing are among the reasons that facilitate. Patients experience severe pain in the first step they take after sitting for a long time or when they get up in the morning and start to walk and the pain is triggered by the tension of the plantar fascia and overlapping weight onto the foot. A large number of conservative methods have been used in the treatment of plantar fasciitis. Anti-inflammatory agents (Non-steroidal anti-inflammatory drugs, steroid injections), physical therapy modalities (iontophoresis, ultrasound, extracorporeal shock wave therapy, electrical stimulation, cryotherapy, and whirlpool), manual therapy, stretching therapy and external support (orthosis and banding) treatment most of these methods. Orthosis and taping aim to correct poor biomechanics in the foot while most of the other treatment programs are suppressing symptoms. Extracorporeal shock wave therapy (ESWT), which is another treatment modality that is used effectively in treatment, is currently preferred in delayed and nonunion fractures, calcified tendinitis of the shoulder, lateral epicondylitis, plantar fasciitis, patellar tendinitis, and calcaneal spur. In a recent prospective study, ESWT treatment was not superior to Kinesio-taping, and both treatments were found to be similar in both pain reduction and increased functionality.

ELIGIBILITY:
Inclusion Criteria:

* Pain when the plantar fascia is palpated,
* Imaging of calcaneal spur radiographically,
* Description of the first step pain, after prolonged resting or awakening in the morning
* Continue with pain despite other conservative methods (NSAI, exercise, etc.)

Exclusion Criteria:

* History of steroid injection in the heel region for the same diagnosis in the last three months,
* Rheumatic disease,
* Coagulopathy, thrombophlebitis, neoplasia, systemic inflammatory diseases,
* Foot and or lumbar surgery, symptoms of lumbar radiculopathy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2019-08-05 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Visual analog scale | 30 days
  Pain on the plantar heel were evaluated with the visual analog scale (0-10 mm). High scores indicate increased pain.

SECONDARY OUTCOMES:
Heel tenderness index | 30 days
  Evaluation of the sensitivity of the heel by the physician (Heel tenderness index: 0= no pain, 1= painful, 2= painful and winces and 3= painful, winces and withdraws).
Foot function index | 30 days
  It measures the impact of foot pathology on function in terms of pain, disability and activity restriction. The questionnaire consists of 23 self-reported items divided into 3 subscales on the basis of patient values: pain, disability and activity limitation.

CONTACTS AND LOCATIONS:
Overall Officials: Yeliz Bahar Ozdemir, Principal Investigator — Hitit University Erol Olcok Training and Research Hospital
Locations (1):
- Hitit University Erol Olcok Training and Research Hospital, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: 60 days

REFERENCES:
- [Background] Frassanito P, Cavalieri C, Maestri R, Felicetti G. Effectiveness of Extracorporeal Shock Wave Therapy and kinesio taping in calcific tendinopathy of the shoulder: a randomized controlled trial. Eur J Phys Rehabil Med. 2018 Jun;54(3):333-340. doi: 10.23736/S1973-9087.17.04749-9. Epub 2017 Nov 29. PMID 29185674
- [Background] Ordahan B, Turkoglu G, Karahan AY, Akkurt HE. Extracorporeal Shockwave Therapy Versus Kinesiology Taping in the Management of Plantar Fasciitis: A Randomized Clinical Trial. Arch Rheumatol. 2017 Apr 17;32(3):227-233. doi: 10.5606/ArchRheumatol.2017.6059. eCollection 2017 Sep. PMID 30375530
- [Background] Zielinski J. [Treatment of uterine corpus cancer of the I/1 stage. I. Complex treatment of uterine corpus cancer]. Ginekol Pol. 1975 Jan;46(1):49-55. No abstract available. Polish. PMID 1110027
- [Background] Kuyucu E, Gulenc B, Bicer H, Erdil M. Assessment of the kinesiotherapy's efficacy in male athletes with calcaneal apophysitis. J Orthop Surg Res. 2017 Oct 6;12(1):146. doi: 10.1186/s13018-017-0637-5. PMID 28985751
- [Derived] Bahar-Ozdemir Y, Atan T. Effects of adjuvant low-dye Kinesio taping, adjuvant sham taping, or extracorporeal shockwave therapy alone in plantar fasciitis: A randomised double-blind controlled trial. Int J Clin Pract. 2021 May;75(5):e13993. doi: 10.1111/ijcp.13993. Epub 2021 Jan 21. PMID 33410228